CLINICAL TRIAL: NCT06471868
Title: An Open-label, Randomized, Multiple-dose, 2-sequence, 2-period, Crossover, Phase 1 Clinical Trial to Evaluate the Safety and the Pharmacokinetics of IY-HCR21 Compared to IY-MIC in Healthy Adult Volunteers
Brief Title: Study to Evaluate Pharmacokinetic and Pharmacodynamic Drug Interactions and Safety of IY-HCR21 and IY-MIC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IY-HTBC01
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Pharmacokinetics
Keywords: a parasympathomimetic choline carbamate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group (Active Comparator): Period 1 : IY-HCR21 1Tab, BID
  Period 2 : IY-MIC 1Tab, QID
  Interventions: Drug: IY-HCR21; Drug: IY-MIC
- B group (Active Comparator): Period 1 : IY-MIC 1Tab, QID
  Period 2 : IY-HCR21 1Tab, BID
  Interventions: Drug: IY-HCR21; Drug: IY-MIC

INTERVENTIONS:
Drug: IY-HCR21 — Betanechol 50mg
Drug: IY-MIC — Betanechol 25mg

SUMMARY:
This study evaluate the pharmacokinetic and safety of IY-HCR21

DETAILED DESCRIPTION:
Phase 1 study to evaluate the safety and the pharmacokinetics of IY-HCR21 in healthy adult volunteers under multiple-dose condition

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers aged 19 years and above at screening
2. A volunteer who weighs ≥ 50kg (≥ 45kg for women) and has a body mass index(BMI)* of ≥18.0 and ≤ 30 at screening

   *BMI(body mass index, kg/m^2)= Body weight (kg)/[height (m)^2]
3. No clinically significant congenital or treatment-requiring chronic medical conditions and no pathological symptoms or findings on internal medicine examination (including EEG, electrocardiogram, thoracic and gastroscopy or gastrointestinal radiology, if necessary)
4. A person who is determined by the principal investigator (or a physician delegated by the principal investigator) to be suitable as a patient as a result of diagnostic tests (e.g., haematology, blood chemistry, serology, urinalysis) and electrocardiograms (ECG) set and conducted according to the characteristics of the investigational drug at the time of screening.
5. Agree that they or their spouse or partner is using a medically accepted method of contraception* (but not hormonal agents) to exclude the possibility of pregnancy from the date of the first dose of investigational drug until 7 days after the last dose of investigational drug, and agree not to provide sperm or eggs
6. Signed the consent form freely and voluntarily after being fully informed and understanding the purpose, content, characteristics of the investigational drug, and expected adverse events of this study.

Exclusion Criteria:

1. Have taken drugs that induce or inhibit drug metabolising enzymes, such as barbiturates, within 30 days prior to study entry (first dose day) or have taken drugs that may interfere with this study within 10 days prior to study entry (first dose day)
2. Participated in a bioequivalence study or other clinical trial within 6 months prior to study initiation (first dose) and received an investigational product
3. blood donation within 8 weeks prior to study entry (first dose day) or component donation within 2 weeks
4. Have a history of gastrointestinal surgery (except appendectomy and hernia surgery) that may affect the absorption of the drug
5. Excessive alcohol consumption within 1 month prior to study entry (first dose day)
6. Patients with any of the following conditions

   * Patients with mechanical obstruction of the gastrointestinal tract or urinary tract
   * spastic gastrointestinal diseases, stomach ulcers, acute inflammatory diseases of the gastrointestinal tract
   * Patients with peritonitis
   * Patients with vasovagal dystonia
   * Patients with asthma
   * Patients with hyperthyroidism
   * Patients with coronary artery occlusion
   * Bradycardia, atrioventricular conduction disorder, vasomotor instability
   * Hypotension, hypertension
   * Patients with myocardial infarction, severe heart disease
   * Patients with epilepsy and parkinsonism
   * Patients treated with anticholinesterase agents
   * Patients with unhealed gastrointestinal anastomoses
   * Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
   * Patients who are hypersensitive to or have a history of allergy to Yellow No. 4 (tartrazine)
   * Patients with a history of hypersensitivity to any of the main ingredients or excipients of this medicine
7. Have a history of clinically significant psychiatric disorders
8. For reasons other than the above inclusion/exclusion criteria, the principal investigator (or delegated investigator) deems the subject unsuitable for this study.
9. For female volunteers, suspected pregnancy or lactation

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-06-25 (Estimated); Study Completion 2024-07-02 (Estimated)

PRIMARY OUTCOMES:
Betanechol AUCt,ss | Day 1 : Predose(0 hour), Day 2 : Predose(0 hour) Day 3 : Predose(0 hour), Afterdose (0.5, 1, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 12.5, 13, 13.5, 14, 14.5, 15, 16, 16.5, 17, 18, 18.5, 19, 19.5, 20, 20.5, 21, 22, 24, 36, 48)
  Betanechol AUCt,ss(Area under the plasma drug concentration-time curve in steady state)
Betanechol Cmax,ss | Day 1 : Predose(0 hour), Day 2 : Predose(0 hour) Day 3 : Predose(0 hour), Afterdose (0.5, 1, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 12.5, 13, 13.5, 14, 14.5, 15, 16, 16.5, 17, 18, 18.5, 19, 19.5, 20, 20.5, 21, 22, 24, 36, 48)
  Betanechol Cmax,ss (Maximum plasma concentration in steady state)

SECONDARY OUTCOMES:
AUCinf | Day 1 : Predose(0 hour), Day 2 : Predose(0 hour) Day 3 : Predose(0 hour), Afterdose (0.5, 1, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 12.5, 13, 13.5, 14, 14.5, 15, 16, 16.5, 17, 18, 18.5, 19, 19.5, 20, 20.5, 21, 22, 24, 36, 48)
  Betanechol AUCinf(Area under the plasma drug concentration-time curve from time 0 to infinity)
t1/2 | Day 1 : Predose(0 hour), Day 2 : Predose(0 hour) Day 3 : Predose(0 hour), Afterdose (0.5, 1, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 12.5, 13, 13.5, 14, 14.5, 15, 16, 16.5, 17, 18, 18.5, 19, 19.5, 20, 20.5, 21, 22, 24, 36, 48)
  Betanechol t1/2(Terminal half-life)
Tmax,ss | Day 1 : Predose(0 hour), Day 2 : Predose(0 hour) Day 3 : Predose(0 hour), Afterdose (0.5, 1, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 12.5, 13, 13.5, 14, 14.5, 15, 16, 16.5, 17, 18, 18.5, 19, 19.5, 20, 20.5, 21, 22, 24, 36, 48)
  Betanechol Tmax,ss(Time to maximum plasma concentration in steady state)
AUCt/AUCinf | Day 1 : Predose(0 hour), Day 2 : Predose(0 hour) Day 3 : Predose(0 hour), Afterdose (0.5, 1, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 12.5, 13, 13.5, 14, 14.5, 15, 16, 16.5, 17, 18, 18.5, 19, 19.5, 20, 20.5, 21, 22, 24, 36, 48)
  Betanechol AUCt/AUCinf
AUC24 | Day 1 : Predose(0 hour), Day 2 : Predose(0 hour) Day 3 : Predose(0 hour), Afterdose (0.5, 1, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 12.5, 13, 13.5, 14, 14.5, 15, 16, 16.5, 17, 18, 18.5, 19, 19.5, 20, 20.5, 21, 22, 24)
  Betanechol AUC24 (Area Under the Plasma Concentration-Time curve in 24hour)
Cmin,ss | Day 1 : Predose(0 hour), Day 2 : Predose(0 hour) Day 3 : Predose(0 hour), Afterdose (0.5, 1, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 12.5, 13, 13.5, 14, 14.5, 15, 16, 16.5, 17, 18, 18.5, 19, 19.5, 20, 20.5, 21, 22, 24, 36, 48)
  Betanechol Cmin,ss (Minimum plasma concentration in steady state)

CONTACTS AND LOCATIONS:
Overall Officials: Seung Hyun Kang, MD, PhD, Study Director — H Plus Yangji Hospital
Locations (1):
- H plus Yangji Hospital, Seoul, Gwanak-gu, South Korea